CLINICAL TRIAL: NCT02953847
Title: The Bioavailability of Rifampicin in Fixed Dose Combinations (FDCs) Widely Used in South Africa to Treat Drug-susceptible Tuberculosis (TB)
Brief Title: The Bioavailability of Rifampicin in (FDCs) Widely Used in South Africa to Treat Drug-susceptible (TB)
Acronym: BIO3FDC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Helen Margaret McIlleron, Senior Research Officer, University of Cape Town
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BIO3FDC
Record Dates: First submitted 2016-09-05; First posted 2016-11-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- sequence 1 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75
- sequence 2 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75
- sequence 3 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75
- sequence 4 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75
- sequence 5 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75
- sequence 6 (Other): Rifafour e-275®, Sanofi-Aventis /Rimactazid 150/75, Sandoz/ Rimactane® 150 mg capsules, Sandoz
  - 24 healthy volunteers will receive single doses of the 3 rifampicin containing products with a washout of 14 days between doses. Each volunteer will be randomised to receive the 3 doses in one of 6 sequences
  Interventions: Drug: Rimactane; Drug: Rifafour e-275; Drug: Rimactazid 150/75

INTERVENTIONS:
Drug: Rimactane — 150 mg capsules, Sandoz MCC registration # A/20.2.3/784
  Other Names: Rifampicin
Drug: Rifafour e-275 — Rifampicin/isoniazid/pyrazinamide/ethambutol 150/75/400/275 mg This 4-drug FDC is the most widely used 4-drug FDC in South Africa with an estimated 100% of the SA DOH tender.
Drug: Rimactazid 150/75 — Rifampicin/isoniazid 150/75 mg This 2-drug FDC is one of 2 widely used 2-drug FDCs in South Africa, with an estimated 30% of the SA DOH tender. Rifinah® made by Sanofi-Aventis holds about 70% of the tender, however as the Sanofi-Aventis 4-drug FDC will also be evaluated.
  Other Names: Rifampicin / Isoniazid

SUMMARY:
3-way cross-over single dose design evaluating bioavailability of 2 rifampicin-containing FDCs vs a single drug comparator in healthy volunteers

DETAILED DESCRIPTION:
In this study the 4- and 2-drug FDCs (for intensive and continuation phases respectively) widely used within the South African treatment program will be evaluated in a comparative bioavailability study against a single drug rifampicin product registered by the South African Medicines Control Council. A three-way, single dose, cross-over study will be conducted in 24 healthy volunteers

ELIGIBILITY:
Inclusion

* You need to be between the ages of 18-55 years
* Have a Body mass index (BMI) of 19-30 kg/m2
* Weigh 45 kg or more
* Be a non-smoker
* Be found to be in normal health on history and examination
* To have normal blood and urine test results
* If you are a woman of child-bearing age, you need to be prepared to not have sexual intercourse, or use a safe form of contraception, until the end of the study

Exclusion

* You are unable to fully understand and comply with the study procedures, requirements and time commitments.
* Are currently enrolled in any other study evaluating drugs, biologics or devices
* You have TB, or have had TB before
* You abuse or have abused drugs or alcohol
* You have, or have had, drug allergy, severe asthma, or active or recurrent allergic disease
* You are pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Cmax | 1 year

OTHER OUTCOMES:
AUC to 12 h | 1 year
AUC to infinity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen M McIlleron, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes